CLINICAL TRIAL: NCT00720304
Title: A Phase II Study of the Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor, Erlotinib, in Combination With Docetaxel and Radiation in Locally Advanced Squamous Cell Cancer of the Head and Neck
Brief Title: Erlotinib, Docetaxel, and Radiation Therapy in Stage III or Stage IV Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5307
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Erlotinib Hydrochloride; In Situ Hybridization, Fluorescence; Polymerase Chain Reaction; Immunoenzyme Techniques; Immunohistochemistry; Radiotherapy, Intensity-Modulated; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- oral erlotinib hydrochloride (Experimental)
  Interventions: Drug: docetaxel; Drug: erlotinib hydrochloride; Genetic: fluorescence in situ hybridization; Genetic: polymerase chain reaction; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: therapeutic conventional surgery; Radiation: intensity-modulated radiation therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: docetaxel — Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
Drug: erlotinib hydrochloride — oral erlotinib hydrochloride once daily for up to 2 years in the absence of disease progression or unacceptable toxicity
Genetic: fluorescence in situ hybridization — Patients undergo blood sample, tissue biopsy, mucosal scraping, and saliva collection at baseline and periodically during study. Samples are analyzed for markers of angiogenic activity (VEGF, sVEGFR-2, sKIT, ICAM, and PDGF), pharmacokinetic studies, gene expression profile, and human papilloma virus DNA by enzyme linked immunosorbent assay (ELISA), immunohistochemistry, fluorescence in situ hybridization (FISH), and PCR.
Genetic: polymerase chain reaction — Patients undergo blood sample, tissue biopsy, mucosal scraping, and saliva collection at baseline and periodically during study. Samples are analyzed for markers of angiogenic activity (VEGF, sVEGFR-2, sKIT, ICAM, and PDGF), pharmacokinetic studies, gene expression profile, and human papilloma virus DNA by enzyme linked immunosorbent assay (ELISA), immunohistochemistry, fluorescence in situ hybridization (FISH), and PCR.
Other: immunoenzyme technique — Patients undergo blood sample, tissue biopsy, mucosal scraping, and saliva collection at baseline and periodically during study. Samples are analyzed for markers of angiogenic activity (VEGF, sVEGFR-2, sKIT, ICAM, and PDGF), pharmacokinetic studies, gene expression profile, and human papilloma virus DNA by enzyme linked immunosorbent assay (ELISA), immunohistochemistry, fluorescence in situ hybridization (FISH), and PCR.
Other: immunohistochemistry staining method — Patients undergo blood sample, tissue biopsy, mucosal scraping, and saliva collection at baseline and periodically during study. Samples are analyzed for markers of angiogenic activity (VEGF, sVEGFR-2, sKIT, ICAM, and PDGF), pharmacokinetic studies, gene expression profile, and human papilloma virus DNA by enzyme linked immunosorbent assay (ELISA), immunohistochemistry, fluorescence in situ hybridization (FISH), and PCR.
Other: laboratory biomarker analysis — Patients undergo blood sample, tissue biopsy, mucosal scraping, and saliva collection at baseline and periodically during study. Samples are analyzed for markers of angiogenic activity (VEGF, sVEGFR-2, sKIT, ICAM, and PDGF), pharmacokinetic studies, gene expression profile, and human papilloma virus DNA by enzyme linked immunosorbent assay (ELISA), immunohistochemistry, fluorescence in situ hybridization (FISH), and PCR.
Other: pharmacological study — Patients undergo blood sample, tissue biopsy, mucosal scraping, and saliva collection at baseline and periodically during study. Samples are analyzed for markers of angiogenic activity (VEGF, sVEGFR-2, sKIT, ICAM, and PDGF), pharmacokinetic studies, gene expression profile, and human papilloma virus DNA by enzyme linked immunosorbent assay (ELISA), immunohistochemistry, fluorescence in situ hybridization (FISH), and PCR.
Procedure: therapeutic conventional surgery — At 6-8 weeks after completion of chemoradiotherapy, patients with N2 or greater cervical lymph node involvement at baseline or with residual disease may undergo surgery.Patients with persistent disease during study therapy undergo salvage surgery 6-12 weeks after completion of chemoradiotherapy.
Radiation: intensity-modulated radiation therapy — radiotherapy (may be intensity-modulated) once daily for 8 weeks in the absence of disease progression or unacceptable toxicity.
Radiation: radiation therapy — radiotherapy (may be intensity-modulated) once daily for 8 weeks in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving erlotinib together with docetaxel and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well erlotinib given together with docetaxel and radiation therapy works in treating patients with stage III or stage IV squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with locally advanced squamous cell carcinoma of the head and neck treated with erlotinib hydrochloride in combination with docetaxel and radiotherapy.

Secondary

* Determine objective response rate, locoregional control rate, duration of response, patterns of failure, and overall survival in patients treated with this regimen.
* Determine the toxicities of this regimen in these patients.
* Determine the dose and effect of this treatment on biologic correlates in tumor tissue and/or surrounding mucosa.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib hydrochloride once daily for up to 2 years in the absence of disease progression or unacceptable toxicity. Beginning on week 3, patients receive docetaxel IV over 1 hour once a week and radiotherapy (may be intensity-modulated) once daily for 8 weeks in the absence of disease progression or unacceptable toxicity.

At 6-8 weeks after completion of chemoradiotherapy, patients with N2 or greater cervical lymph node involvement at baseline or with residual disease may undergo surgery. Patients with persistent disease during study therapy undergo salvage surgery 6-12 weeks after completion of chemoradiotherapy.

Patients undergo blood sample, tissue biopsy, mucosal scraping, and saliva collection at baseline and periodically during study. Samples are analyzed for markers of angiogenic activity (VEGF, sVEGFR-2, sKIT, ICAM, and PDGF), pharmacokinetic studies, gene expression profile, and human papilloma virus DNA by enzyme linked immunosorbent assay (ELISA), immunohistochemistry, fluorescence in situ hybridization (FISH), and PCR.

After completion of study therapy, patients will be evaluated every 4-8 weeks for 1 year, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 2 years, and then once a year thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced squamous cell carcinoma of the head and neck

  * Stage III or IV disease

    * No distant metastatic disease
* Measurable disease (according to RECIST)
* No salivary gland and paranasal sinus squamous cell carcinoma
* No known brain metastases or direct cerebral invasion by tumor

  * Intracranial extension (without cerebral involvement) may be allowed

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥10 g/dL
* Total bilirubin normal
* Alkaline phosphatase AND AST and ALT meeting the following criteria:

  * Alkaline phosphatase normal AND AST and ALT ≤ 5 times upper limit of normal (ULN)
  * Alkaline phosphatase ≤ 2.5 times ULN AND AST and ALT ≤ 2.5 times ULN
  * Alkaline phosphatase ≤ 5 times ULN AND AST and ALT normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* No clinically significant heart disease including any of the following:

  * NYHA class III or IV heart disease
  * Significant arrhythmias requiring medication
  * Symptomatic coronary artery disease
  * Myocardial infarction within the previous six months
  * Second- or third-degree heart block or bundle-branch block
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after completion of study therapy
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib hydrochloride or docetaxel, including other drugs formulated with polysorbate 80
* No pre-existing peripheral neuropathy ≥ grade 2
* No uncontrolled concurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would preclude compliance with study requirements
* No HIV positivity
* No other prior malignancy except for any of the following:

  * Squamous cell or basal cell carcinoma of the skin
  * Carcinoma in situ of the cervix
  * Cancer that was treated more than 5 years ago and the patient has remained disease-free
* Not poorly compliant

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or investigational antitumor drug
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-11-19 (Actual); Primary Completion 2015-11-13 (Actual); Study Completion 2015-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min Yao, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CASE5307 - Oral Erlotinib Hydrochloride: Weekly docetaxel (20 mg/m2), EGF-R inhibition: Erlotinib 150 mg/day (prior to, during and up to two years following XRT)
- Participants From CWRU1301: Participants from CWRU1301 - NCT00049283 who received Docetaxel 20 mg/m2/wk Erlotinib 150 mg/day XRT
Period: Overall Study
Arm/Group | CASE5307 - Oral Erlotinib Hydrochloride | Participants From CWRU1301
Started | 37 | 6
Completed | 8 | 1
Not Completed | 29 | 5
Not completed — Withdrawal by Subject | 14 | 1
Not completed — Death | 1 | 0
Not completed — Physician Decision | 5 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Disease progression | 6 | 1

BASELINE CHARACTERISTICS:
Population: 37 participants enrolled on CASE5307 (NCT00720304), 6 participants enrolled on CWRU1301 (NCT00049283)
Groups:
- CASE5307 - Oral Erlotinib Hydrochloride: Docetaxel, erlotinib hydrochloride, fluorescence in situ hybridization, polymerase chain reaction, immunoenzyme technique, immunohistochemistry staining method, laboratory biomarker analysis, pharmacological study, therapeutic conventional surgery, intensity-modulated radiation therapy, radiation therapy
- Total: Total of all reporting groups
Arm/Group | CASE5307 - Oral Erlotinib Hydrochloride | Participants From CWRU1301 | Total
Number analyzed (Participants) | 37 | 6 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 6 | 31
  >=65 years | 12 | 0 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 28 | 5 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 5 | 40
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 32 | 3 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 37 | 6 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Disease-Free Survival (DFS) at 3 Years
Description: Percent of participants with Disease-Free survival (DFS) at 3 years. Assessed from date of treatment to date of death or date of disease progression, and to date of last follow-up for those still alive and progression free. Disease-free Survival percentages were calculated using Kaplan-Meier estimates.
Time Frame: 3 yrs after treatment
Population: Participants enrolled in study
Measure: Number; unit: Percent
Arm/Group | Oral Erlotinib Hydrochloride
Number analyzed (Participants) | 43
Percent | 69.5

2. Primary Outcome: Time to Progression (TTP)
Description: Time from start of treatment to first documented occurrence of progressive disease (PD). PD defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 3 yrs after treatment
Population: Data not available because response data not collected
Groups:
- Oral Erlotinib Hydrochloride: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
  erlotinib hydrochloride: oral erlotinib hydrochloride once daily for up to 2 years in the absence of disease progression or unacceptable toxicity
  fluorescence in situ hybridization: Patients undergo blood sample, tissue biopsy, mucosal scraping, and saliva collection at baseline and periodically during study. Samples are analyzed for markers of angiogenic activity (VEGF, sVEGFR-2, sKIT, ICAM, and PDGF), pharmacokinetic studies, gene expression profile, and human papilloma virus DNA by enzyme linked immunosorbent assay (ELISA), immunohistochemistry, fluorescence in situ hybridization (FISH), and PCR.
  polymerase chain reaction: Patients undergo blood sample, tissue biopsy, mucosal scraping, and saliva collection at baseline and periodically during study. Samples are analyzed for markers of angiogenic activity (VEGF, sVEGFR-2, sKIT, ICAM, and PDGF), pharmacokinetic studies, gene expression profi
Arm/Group | Oral Erlotinib Hydrochloride
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Rate (Complete Response, Partial Response, Stable Disease, and Disease Progression)
Description: Response rate according to response criteria, which defines the following:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 3 yrs after treatment
Population: Data not available because response data not collected
Arm/Group | Oral Erlotinib Hydrochloride
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Percent of participants alive at follow-up time. Overall survival time is evaluated from the date of treatment to date of death, and to date of last follow-up for those still alive.
Time Frame: 3 years
Population: Participants enrolled in study
Measure: Number; unit: Percent
Arm/Group | Oral Erlotinib Hydrochloride
Number analyzed (Participants) | 43
Percent | 81

5. Secondary Outcome: Number of Participants With Acute Grade III/IV Treatment-related Toxicities
Description: Number of participants with acute grade III/IV treatment-related toxicities
Time Frame: evaluated every 2 weeks, up to 3 years
Population: Participants enrolled in study
Measure: Count of Participants; unit: Participants
Groups:
- Lymphopenia: Lymphopenia
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
- Neutropenia: Neutropenia
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
- Anemia: Anemia
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
- Oral Mucositis: Oral mucositis
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
- Radiation Dermatitis: Radiation dermatitis
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
- Acneiform Skin Rash: Acneiform skin rash
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
- Dysphagia: Dysphagia
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
- Anorexia: Anorexia
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
- Nausia/Vomiting: Nausia/vomiting
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
- Dehydration: Dehydration
  Participant intervention: docetaxel: Beginning on week 3, patients receive docetaxel IV over 1 hour once a week
Arm/Group | Lymphopenia | Neutropenia | Anemia | Oral Mucositis | Radiation Dermatitis | Acneiform Skin Rash | Dysphagia | Anorexia | Nausia/Vomiting | Dehydration
Number analyzed (Participants) | 43 | 43 | 43 | 43 | 43 | 43 | 43 | 43 | 43 | 43
Participants
  Grade 3 | 24 | 2 | 3 | 14 | 15 | 4 | 20 | 13 | 7 | 2
  grade 4 | 17 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0

6. Secondary Outcome: Percent of Participants With Local Failure-free Survival
Description: Participants with Local absence of relapse or recurrence or progression within the prescribed radiation field.
Time Frame: At 3 years
Population: Participants enrolled in study
Measure: Number; unit: percent
Arm/Group | Oral Erlotinib Hydrochloride
Number analyzed (Participants) | 43
percent | 90

7. Other Pre Specified Outcome: Predictive Values of EGFR/TGF-α, VEGF
Time Frame: collection at baseline and periodically during study.
Reporting Status: Not Posted

8. Secondary Outcome: Percent of Participants With Regional Failure-free Survival
Description: Participants with the regional absence of relapse or recurrence or progression within the prescribed radiation field. Failure-free Survival percentages were calculated using Kaplan-Meier estimates.
Time Frame: At 3 years
Population: Participants enrolled in study
Measure: Number; unit: percent (Kaplan-Meier estimates)
Arm/Group | Oral Erlotinib Hydrochloride
Number analyzed (Participants) | 43
percent (Kaplan-Meier estimates) | 87.1

9. Secondary Outcome: Percent of Participants With Locoregional Failure-free Survival
Description: Participants with the locoregional absence of relapse or recurrence or progression within the prescribed radiation field. Locoregional failure-free survival percentages were calculated using Kaplan-Meier estimates.
Time Frame: At 3 years
Population: Participants enrolled in study
Measure: Number; unit: percent (Kaplan-Meier estimates)
Arm/Group | Oral Erlotinib Hydrochloride
Number analyzed (Participants) | 43
percent (Kaplan-Meier estimates) | 82.4

10. Secondary Outcome: Percent of Participants With Distant Metastasis-free Survival
Description: Percent of participants with distant metastasis-free survival
Time Frame: At 3 years
Population: Participants enrolled in study
Measure: Number; unit: percent
Arm/Group | Oral Erlotinib Hydrochloride
Number analyzed (Participants) | 43
percent | 83.7

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Toxicity assessment performed at baseline, every two weeks until week 10, and then monthly until off-study (up to 3 years)
Groups:
- Oral Erlotinib Hydrochloride: Docetaxel, erlotinib hydrochloride, fluorescence in situ hybridization, polymerase chain reaction, immunoenzyme technique, immunohistochemistry staining method, laboratory biomarker analysis, pharmacological study, therapeutic conventional surgery, intensity-modulated radiation therapy, radiation therapy
Arm/Group | Oral Erlotinib Hydrochloride | Participants From CWRU1301
All-Cause Mortality (participants affected / at risk) | 11/37 | 4/6
Serious Adverse Events (participants affected / at risk) | 11/37 | 1/6
Other Adverse Events (participants affected / at risk) | 33/37 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Erlotinib Hydrochloride (N=37) | Participants From CWRU1301 (N=6)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4 (4) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hemorrhage, GI - Lower GI (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 2 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rash: dermatitis associated with radiation - Radiation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Valvular heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Peripheral arterial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Erlotinib Hydrochloride (N=37) | Participants From CWRU1301 (N=6)
Hemoglobin (Blood and lymphatic system disorders) | 32 (125) | 5 (33)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 5 (7) | 0 (0)
Pain - External ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain - Eye (Ear and labyrinth disorders) | 1 (3) | 0 (0)
Pain - Middle ear (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Auditory congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Auditory blockage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 2 (2) | 0 (0)
Endocrine - increased TSH (Endocrine disorders) | 1 (1) | 0 (0)
Ocular/Visual nonblood (Eye disorders) | 1 (1) | 0 (0)
Itching eyes (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (26) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 16 (44) | 4 (12)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 23 (34) | 4 (5)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 33 (109) | 6 (20)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 16 (31) | 2 (3)
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 30 (119) | 0 (0)
Nausea (Gastrointestinal disorders) | 25 (55) | 3 (4)
Pain - Abdomen (Gastrointestinal disorders) | 14 (17) | 0 (0)
Pain - Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain - Lip (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain - Oral cavity (Gastrointestinal disorders) | 22 (54) | 1 (1)
Pain - Stomach (Gastrointestinal disorders) | 1 (1) | 1 (1)
Salivary gland changes/saliva (Gastrointestinal disorders) | 23 (59) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (36) | 2 (2)
Pain - oral cavity, throat (Gastrointestinal disorders) | 1 (3) | 0 (0)
Hemorrhage/Bleeding - PEG site (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain associated with swallowing and coughing (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain - tongue (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain - eipgastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain - mouth and throat (Gastrointestinal disorders) | 1 (4) | 2 (5)
Edema (General disorders) | 0 (0) | 4 (5)
Edema: head and neck (General disorders) | 6 (6) | 0 (0)
Edema: limb (General disorders) | 4 (4) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 33 (103) | 6 (19)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 7 (12) | 3 (3)
Pain - Face (General disorders) | 9 (10) | 1 (1)
Rigors/chills (General disorders) | 9 (11) | 2 (2)
Constitutional Symptoms - nonblood (General disorders) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Cytokine release syndrome/acute infusion reaction (Immune system disorders) | 1 (6) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Abdomen NOS (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Eye NOS (Infections and infestations) | 1 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Neck NOS (Infections and infestations) | 2 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Nerve-peripheral (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Oral cavity-gums (gingivitis) (Infections and infestations) | 5 (5) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Paranasal (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 5 (5) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection - thrush (Infections and infestations) | 2 (2) | 0 (0)
Infection - clostridium diff. (Infections and infestations) | 1 (1) | 0 (0)
Infection - nonblood (Infections and infestations) | 1 (1) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rash: dermatitis associated with radiation - Chemoradiation (Injury, poisoning and procedural complications) | 29 (89) | 0 (0)
Rash: dermatitis associated with radiation - Radiation (Injury, poisoning and procedural complications) | 4 (7) | 1 (1)
Alkaline phosphatase (Investigations) | 10 (27) | 2 (6)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 16 (32) | 3 (5)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 12 (31) | 4 (12)
Bilirubin (hyperbilirubinemia) (Investigations) | 15 (47) | 3 (8)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 1 (1) | 0 (0)
Creatinine (Investigations) | 8 (11) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 4 (14) | 0 (0)
Leukocytes (total WBC) (Investigations) | 19 (89) | 4 (19)
Lymphopenia (Investigations) | 33 (328) | 4 (32)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 (8) | 1 (1)
Platelets (Investigations) | 8 (25) | 1 (10)
PTT (Partial Thromboplastin Time) (Investigations) | 1 (3) | 0 (0)
Weight loss (Investigations) | 30 (84) | 6 (7)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 31 (121) | 4 (16)
Anorexia (Metabolism and nutrition disorders) | 28 (80) | 5 (13)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 21 (64) | 4 (14)
Dehydration (Metabolism and nutrition disorders) | 13 (18) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 19 (97) | 5 (32)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 6 (11) | 3 (11)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 23 (43) | 4 (4)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 10 (12) | 1 (6)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 16 (37) | 3 (4)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 13 (25) | 1 (4)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 6 (7) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 29 (86) | 2 (8)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Bone growth: spine kyphosis/lordosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4)
Pain - Back (Musculoskeletal and connective tissue disorders) | 10 (14) | 0 (0)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 5 (8) | 0 (0)
Pain - Chest/thorax (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 5 (9) | 0 (0)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - Neck (Musculoskeletal and connective tissue disorders) | 13 (22) | 3 (4)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Trismus (difficulty, restriction or pain when opening mouth) (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (5) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 4 (6)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (2) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 3 (4) | 2 (4)
Pain - Head/headache (Nervous system disorders) | 6 (10) | 1 (1)
Pain - Sinus (Nervous system disorders) | 1 (1) | 0 (0)
Taste alteration (dysgeusia) (Nervous system disorders) | 17 (45) | 3 (7)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 20 (44) | 1 (1)
Mood alteration - Agitation (Psychiatric disorders) | 6 (8) | 0 (0)
Mood alteration - Anxiety (Psychiatric disorders) | 11 (16) | 1 (2)
Mood alteration - Depression (Psychiatric disorders) | 9 (14) | 0 (0)
Personality/behavioral (Psychiatric disorders) | 1 (2) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pain - Kidney (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (28) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (15) | 4 (4)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hemorrhage, pulmonary/upper respiratory - Pharynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Mucositis/stomatitis (clinical exam) - Pharynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstruction/stenosis of airway - Pharynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 27 (78) | 3 (7)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 24 (55) | 2 (4)
Chest tightness during Taxotere infusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased mucous in throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pressure (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thick sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Mucous secretion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (20) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 13 (17) | 3 (3)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain - Scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain - Skin (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 18 (33) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12 (24) | 6 (29)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 26 (91) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Pain - Skin of face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
small lesion on shaft of penis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
sebacous cyst on chest (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 6 (13) | 0 (0)
Hot flashes/flushes (Vascular disorders) | 4 (5) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
unsteady gait (General disorders) | 0 (0) | 1 (1)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
anterior neck irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
sores in nostrils (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dermatitis/erythema neck, ear (open area), lip (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
sores around mouth/lips (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
cracking fingernails (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
face erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
excoriation at trach site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
decubitis ulcer, sacral area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
erythema at PEG tube site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Endocrine-NOS (Endocrine disorders) | 0 (0) | 1 (1)
Mucositis due to radiation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 0 (0) | 6 (29)
ulceration, tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
ulcerated R tonsillar bed (Gastrointestinal disorders) | 0 (0) | 1 (1)
difficulty chewing (Gastrointestinal disorders) | 0 (0) | 1 (1)
early satiety (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Melena/GI bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Infections and infestations) | 0 (0) | 1 (1) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1)
Infection without neutropenia (Infections and infestations) | 0 (0) | 1 (2)
lymphedema, anterior neck (Vascular disorders) | 0 (0) | 1 (1)
Bicarbonate (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
leg cramps at night (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
muscle tightening in back (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (3)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain, R lower quadrant (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
neck achiness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
right neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
right jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
neck/throat pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
pain - R hip and leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain, tracheostomy site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain, PEG tube site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
moderate obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
thick secretions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
nasal drainage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Outcomes data from 6 participants who received the same treatment on CWRU1301 (NCT00049283) were including in the results for this record.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes